CLINICAL TRIAL: NCT00441298
Title: Phase IIb Trial to Assess the Safety and Effectiveness of the Vaginal Microbicide 1% Tenofovir Gel for the Prevention of HIV Infection in Women in South Africa
Brief Title: Safety and Effectiveness Study of a Candidate Vaginal Microbicide for Prevention of HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: FHI 360 (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); CONRAD (Other)
Responsible Party: Principal Investigator, Dr Salim S Abdool Karim, Principal Investigator, Centre for the AIDS Programme of Research in South Africa
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CAPRISA 004; PHSC study #9946
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: HIV Infections
Keywords: microbicides; safety; effectiveness; Tenofovir gel; HIV; young women; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Tenofovir gel (a reverse transcriptase inhibitor)
  Interventions: Drug: Tenofovir gel
- 2 (Placebo Comparator): Universal HEC placebo
  Interventions: Drug: Placebo (Universal HEC placebo)

INTERVENTIONS:
Drug: Tenofovir gel — Participants will be provided with a supply of single-use, pre-filled applicators according to their randomisation. While in the study, participants will be asked to apply a first dose of the assigned study product, 1% tenofovir gel, within 12 hours prior to coitus and insert a second dose as soon as possible within 12 hours after coitus. They will be advised to use only two doses of gel in a 24-hour period.
  Other Names: Tenofovir = Viread
  Arms: 1
Drug: Placebo (Universal HEC placebo) — Participants will be provided with a supply of single-use, pre-filled applicators according to their randomisation. While in the study, participants will be asked to apply a first dose of the assigned study product, placebo gel, within 12 hours prior to coitus and insert a second dose as soon as possible within 12 hours after coitus. They will be advised to use only two doses of gel in a 24-hour period.
  Arms: 2

SUMMARY:
This phase IIb, two-arm, double-blinded, randomised, placebo controlled trial comparing 1% Tenofovir gel with a placebo gel is an expanded safety and effectiveness trial involving 900 young women at risk of sexually transmitted HIV infection. Participants will be provided with a supply of single-use, pre-filled applicators according to their randomisation. While in the study, participants will be asked to apply a first dose of the assigned study gel within 12 hours prior to coitus and insert a second dose as soon as possible within 12 hours after coitus. All participants will receive HIV risk reduction counselling, condoms, and syndromic treatment of sexually transmitted infections, if required.

DETAILED DESCRIPTION:
Purpose: To assess the safety and effectiveness of tenofovir gel, a candidate vaginal microbicide, in sexually active women at risk for human immunodeficiency virus (HIV) infection in South Africa.

Design: Phase IIb, two-arm, double-blind, randomised, controlled trial comparing 1% tenofovir gel with a placebo gel.

Study Population: Sexually active, HIV-uninfected women aged 18 to 40 years in South Africa

Study Size: 900 women

Treatment Regimen: Participants will be provided with a supply of single-use, pre-filled applicators according to their randomisation. While in the study, participants will be asked to apply a first dose of the assigned study product, 1% tenofovir gel or placebo gel, within 12 hours prior to coitus and insert a second dose as soon as possible within 12 hours after coitus. They will be advised to use only two doses of gel in a 24-hour period.

Study Duration: Approximately 30 months in total. Accrual will require approximately 14 months and follow-up will continue until 92 incident HIV infections are observed in the study, which is expected to occur approximately 16 months after the end of the accrual period.

Primary Objective:

To evaluate the effectiveness and safety of a candidate vaginal microbicide, tenofovir gel, when applied intravaginally by women, in preventing sexually transmitted HIV infection.

Secondary Objectives:

* To assess the impact, if any, of tenofovir gel on the incidence rate of deep epithelial disruption
* To assess the impact, if any, of tenofovir gel on viral load in women who become infected with HIV during the trial.
* To assess tenofovir resistance in HIV seroconvertors in the trial
* To ascertain the impact, if any, of tenofovir gel on pregnancy rates and outcomes
* To assess the impact, if any, of product hold at study exit on HIV infection and tenofovir resistance

Ancillary Objective

•To assess the impact, if any, of tenofovir gel in preventing sexually transmitted infections, including herpes simplex virus type 2 (HSV-2) and human papillomavirus (HPV) infections.

Study sites:

* CAPRISA Vulindlela Clinical Research Site, KwaZulu-Natal, South Africa
* CAPRISA eThekwini Clinical Research Site, Durban, South Africa

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years (inclusive)
* Able and willing to provide written informed consent to be screened for, and to enrol in, the study.
* Able and willing to provide adequate locator information for study retention purposes.
* Sexually active, defined as having had vaginal intercourse at least twice in the past 30 days prior to screening.
* HIV negative on testing performed by study staff within 30 days of enrolment.
* Have a negative pregnancy test which was performed by study staff within 21 days of enrolment
* Agree to use a non-barrier form of contraceptive
* Agree to adhere to study visits and procedures

Exclusion Criteria:

* History of adverse reaction to latex.
* Plans any of the following during the next 16 to 30 months (depending the anticipated date of study completion):

  * To travel away from the study site for more than 30 consecutive days.
  * To relocate away from the study site.
  * To become pregnant
  * To enrol in any other study of an investigational product or behaviour modification related to HIV prevention.
* Has a creatinine clearance <50ml/min, as estimated using the method of Cockcroft and Gault(33).
* Has active Hepatitis B infection (since January 2009)
* Has a clinically apparent pelvic examination finding (observed by study staff) involving deep epithelial disruption. Otherwise eligible participants with pelvic examination findings involving deep epithelial disruption may proceed with enrolment after the findings have resolved and the inclusion/exclusion are met.
* Has in the past year participated in any research related to any vaginally applied product/s.
* Has current STI symptoms and/or other reproductive tract infection requiring treatment, as assessed by study staff. Otherwise eligible participants diagnosed during screening with infection(s) requiring treatment may be enrolled provided that treatment has commenced.
* Has any other condition that, based on the opinion of the Investigator or designee, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 889 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change in HIV status compared between arms (tenofovir vs placebo) | Baseline and monthly HIV testing for the duration of the study, an expected average of 18 months
  The effectiveness of tenofovir against HIV infection will be measured by comparing the incidence of HIV in the tenofovir arm with that in the placebo arm

SECONDARY OUTCOMES:
Change in incidence rate of deep epithelial disruption compared between arms | Baseline and monthly assessments for the duration of the study, an expected average of 18 months
  To assess the impact, if any, of tenofovir gel on the incidence rate of deep epithelial disruption
To assess the impact of tenofovir gel on viral load | measured at the first visit post HIV infection, and again 3 months later
  To assess the impact, if any, of tenofovir gel on viral load in women who become infected with HIV during the trial.
To assess tenofovir resistance in HIV seroconvertors in the trial | performed at the post-seroconversion visit
To ascertain the impact, if any, of tenofovir gel on pregnancy rates and outcomes | Assessed at baseline and monthly for the duration of the study, an expected average of 18 months
To assess the impact, if any, of product hold at study exit on HIV infection and tenofovir resistance | Assessed at post study visit
  Assess new HIV seroconversions in the period between study exit and the post study visit (range 2 to 4 months)
Impact of tenofovir gel on other sexually transmitted infections | Change from baseline to study exit
  To assess the impact, if any, of tenofovir gel in preventing sexually transmitted infections, including herpes simplex virus type 2 (HSV-2) and human papillomavirus (HPV) infections

CONTACTS AND LOCATIONS:
Overall Officials: Salim S Abdool karim, MBChB, PhD, Principal Investigator — CAPRISA, University of KwaZulu-Natal; Quarraisha Abdool Karim, PhD, Principal Investigator — CAPRISA, University of KwaZulu-Natal
Locations (2):
- South Africa (2):
  - CAPRISA eThekwini Clinical Research Site, Durban, KwaZulu-Natal
  - CAPRISA, Vulindlela Clinical Research Site, Pietermaritzburg, KwaZulu-Natal

REFERENCES:
- [Background] Mayer KH, Maslankowski LA, Gai F, El-Sadr WM, Justman J, Kwiecien A, Masse B, Eshleman SH, Hendrix C, Morrow K, Rooney JF, Soto-Torres L; HPTN 050 Protocol Team. Safety and tolerability of tenofovir vaginal gel in abstinent and sexually active HIV-infected and uninfected women. AIDS. 2006 Feb 28;20(4):543-51. doi: 10.1097/01.aids.0000210608.70762.c3. PMID 16470118
- [Result] Abdool Karim Q, Abdool Karim SS, Frohlich JA, Grobler AC, Baxter C, Mansoor LE, Kharsany AB, Sibeko S, Mlisana KP, Omar Z, Gengiah TN, Maarschalk S, Arulappan N, Mlotshwa M, Morris L, Taylor D; CAPRISA 004 Trial Group. Effectiveness and safety of tenofovir gel, an antiretroviral microbicide, for the prevention of HIV infection in women. Science. 2010 Sep 3;329(5996):1168-74. doi: 10.1126/science.1193748. Epub 2010 Jul 19. PMID 20643915
- [Derived] Wang Y, Noel-Romas L, Perner M, Knodel S, Molatlhegi R, Hoger S, Birse K, Zuend CF, McKinnon LR, Burgener AD. Non-Lactobacillus-Dominant and Polymicrobial Vaginal Microbiomes Are More Common in Younger South African Women and Predictive of Increased Risk of Human Immunodeficiency Virus Acquisition. Clin Infect Dis. 2023 Apr 17;76(8):1372-1381. doi: 10.1093/cid/ciac938. PMID 36504254
- [Derived] Abdool Karim SS, Abdool Karim Q, Kharsany AB, Baxter C, Grobler AC, Werner L, Kashuba A, Mansoor LE, Samsunder N, Mindel A, Gengiah TN; CAPRISA 004 Trial Group. Tenofovir Gel for the Prevention of Herpes Simplex Virus Type 2 Infection. N Engl J Med. 2015 Aug 6;373(6):530-9. doi: 10.1056/NEJMoa1410649. PMID 26244306
- [Derived] Naranbhai V, Samsunder N, Sandler NG, Roque A, Abdool Karim Q, Ndung'u T, Carr WH, Altfeld M, Douek DC, Abdool Karim SS; CAPRISA 004 Trial Team. Neither microbial translocation nor TLR responsiveness are likely explanations for preexisting immune activation in women who subsequently acquired HIV in CAPRISA 004. J Acquir Immune Defic Syndr. 2013 Jul 1;63(3):294-8. doi: 10.1097/QAI.0b013e31828e604b. PMID 23481666
- [Derived] Matthews LT, Sibeko S, Mansoor LE, Yende-Zuma N, Bangsberg DR, Karim QA. Women with pregnancies had lower adherence to 1% tenofovir vaginal gel as HIV preexposure prophylaxis in CAPRISA 004, a phase IIB randomized-controlled trial. PLoS One. 2013;8(3):e56400. doi: 10.1371/journal.pone.0056400. Epub 2013 Mar 5. PMID 23472071
- [Derived] Naranbhai V, Altfeld M, Abdool Karim Q, Ndung'u T, Abdool Karim SS, Carr WH; Centre for the AIDS Programme of Research in South Africa (CAPRISA) Tenofovir gel Research for AIDS Prevention Science (TRAPS) Team. Natural killer cell function in women at high risk for HIV acquisition: insights from a microbicide trial. AIDS. 2012 Sep 10;26(14):1745-53. doi: 10.1097/QAD.0b013e328357724f. PMID 22781225
- [Derived] Karim QA, Kharsany AB, Frohlich JA, Baxter C, Yende N, Mansoor LE, Mlisana KP, Maarschalk S, Arulappan N, Grobler A, Sibeko S, Omar Z, Gengiah TN, Mlotshwa M, Samsunder N, Karim SS. Recruitment of high risk women for HIV prevention trials: baseline HIV prevalence and sexual behavior in the CAPRISA 004 tenofovir gel trial. Trials. 2011 Mar 7;12:67. doi: 10.1186/1745-6215-12-67. PMID 21385354
- See also: Central website for the Centre for the AIDS Programme of Research in South Africa — http://www.caprisa.org